CLINICAL TRIAL: NCT06583369
Title: The Efficacy and Safety of Liangxue Ointment in the Treatment of Hand-foot Syndrome Caused by VEGFR-TKI Drugs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Lu Si, professor, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022YJZ82
Record Dates: First submitted 2024-09-01; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-04

CONDITIONS: Hand-Foot Syndrome
Keywords: axitinib; Hand-Foot Syndrome; renal cell carcinoma; Melanoma; VEGFR-TKI
MeSH Terms: conditions — Hand-Foot Syndrome; Carcinoma, Renal Cell; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liangxue ointment (Experimental): Apply 2 times a day, 14 days is a course of treatment, and the treatment is 2 courses.
  Interventions: Drug: Liangxue ointment（Traditional Chinese Ointment）
- urea cream (Active Comparator): Apply 2 times a day, 14 days is a course of treatment, and the treatment is 2 courses.
  Interventions: Drug: Urea cream

INTERVENTIONS:
Drug: Liangxue ointment（Traditional Chinese Ointment） — The main ingredients of Liangxue Ointment include: Lithospermum sibiricum, Sanguisorba Sanguis, Rehmannia glutinosa, Gardenia, rhubarb, skullcap, borneol, dragon's blood, olibanum and myrrh.
  Apply 2 times a day, 14 days is a course of treatment, and the treatment is 2 courses.
  Arms: Liangxue ointment
Drug: Urea cream — Apply 2 times a day, 14 days is a course of treatment, and the treatment is 2 courses.
  Arms: urea cream

SUMMARY:
This study was a prospective, single-center randomized controlled trial. The subject of this study is to evaluate the effectiveness and safety of traditional Chinese medicine Liangxue Ointment in the treatment of hand-foot syndrome caused by VEGFR-TKI drugs.

DETAILED DESCRIPTION:
This study was a prospective, single-center randomized controlled trial. Patients with hand-foot syndrome caused by VEGFR-TKI drugs were randomly divided into the experimental group and the control group at a ratio of 1:1 according to the numerical randomization method. All patients are required to avoid inappropriate local friction of hands and feet; avoid heavy physical labor and sun exposure; eat a light diet, avoid spicy and irritating foods, and keep warm. The control group received urea cream application, and the experimental group received Liangxue ointment application.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old, both men and women are welcome;
* Patients with pathologically confirmed malignant tumors;
* Receive treatment with VEGFR-TKI drugs;
* Hand-foot syndrome associated with VEGFR-TKI drugs is judged by the researcher;
* No skin lesions on hands and feet before receiving VEGFR-TKI drug treatment;
* No allergies to the traditional Chinese medicine components of the trial drug;
* Be conscious, have language expression or reading skills, and can communicate normally;
* Estimated survival time ≥3 months;
* ECOG score ≤ 2;
* Ability to comply with the trial protocol, as judged by the investigator;
* Women of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose of the trial drug; men of reproductive potential or women with the possibility of pregnancy must use highly effective contraceptive methods (such as oral contraceptives, oral contraceptives, Intrauterine device, libido control or barrier method combined with spermicide) and continue contraception for 6 months after the end of treatment;
* Voluntarily participate in this clinical trial, understand the research procedures and be able to sign the written informed consent form.

Exclusion Criteria:

* Those with skin ulcers on hands and feet;
* Known allergy to ingredients of Liangxue Ointment;
* Have used other targeted drugs and chemotherapy drugs that cause HFS within 4 weeks;
* Those who have skin lesions on their hands and feet before treatment with VEGFR-TKI drugs or those who have a history of skin diseases;
* Use of medications within 2 weeks that may affect study results (topical antibiotics, topical steroids, and other topical treatments);
* With serious accompanying diseases, such as severe hypertension, diabetes, thyroid disease, heart disease, and mental illness;
* Poor compliance and refusal to cooperate with follow-up visits;
* Other reasons lead the researcher to believe that they are not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-03-25 (Estimated); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
2-week treatment effectiveness | Participants will be followed for an expected average of 4 weeks
  According to the patient's NCI CTCAE grade improvement, it is divided into: 1) The clinical symptoms completely disappear, which is a complete remission; 2) The symptom grade decreases by 1 level or more (not including falling to level 0), which is a partial remission; 3) There is no change in symptoms. , is invalid. Calculate the treatment effectiveness at different time points respectively, and take the 2-week treatment effectiveness as the main research endpoint.

SECONDARY OUTCOMES:
Quality of life improvement value | The quality of life improvement values were calculated each week during treatment, 2 weeks, and 4 weeks after the end of treatment.
  Quality of life improvement value: According to the HFS-14 scale, patients' quality of life scores were scored before and after treatment. Quality of life improvement value = quality of life score before treatment - quality of life score after treatment. The quality of life improvement values were calculated each week during treatment, 2 weeks, and 4 weeks after the end of treatment.
Pain relief rate | Participants will be followed for an expected average of 4 weeks
  Pain relief rate: The NRS numerical scoring method is used to evaluate the pain before and after treatment: 1) The disappearance of pain after treatment is complete relief; 2) The pain score after treatment / the pain score before treatment ≤50% is effective; 3) There is no change in pain, which is invalid. Pain relief rate = (number of complete relief cases + number of effective cases)/total number of cases × 100%.
Drug discontinuation and dose reduction rate | Participants will be followed for an expected average of 4 weeks
  Drug discontinuation and dose reduction: the rate of drug discontinuation or dose reduction in the two groups due to severe hand-foot syndrome caused by VEGFR-TKI drugs.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China